CLINICAL TRIAL: NCT06348290
Title: a Single-center, Non-randomized, Open-label, Self-controlled Phase 1 Clinical Study to Evaluate Drug-drug Interactions of JMKX001899 Tablets in Healthy Subjects
Brief Title: Study to Evaluate the Drug-drug Interaction of JMKX001899 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JY-JM1899-105
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Itraconazole; Midazolam; Rifampin; Dextromethorphan; Rosuvastatin Calcium; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JMKX001899+Itraconazole (Experimental): Enrolled subjects were treated with JMKX001899 on Day 1. Itraconazole was administered orally once daily after a standardized meal from Day 4 to Day 6. JMKX001899 and itraconazole were administered simultaneously after a standardized meal on Day 7. On Day 8 to Day 9, itraconazole was orally administered once after a standard meal
  Interventions: Drug: JMKX001899; Drug: Itraconazole
- JMKX001899+Rifampin (Experimental): Enrolled subjects were treated with JMKX001899 after high fat meal on Day 1 and an empty stomach on Day 4. Rifampin was administered orally once daily on an empty stomac from Day 7 to Day 15, Day 17and Day 18. JMKX001899 and Rigampin were administered simultaneously on an empty stomach on Day 16.
  Interventions: Drug: JMKX001899; Drug: Rifampin
- JMKX001899+Cocktail substrate (Midazolam, dextromethorphan, Rosuvastatin and digoxin) (Experimental): Enrolled subjects were treated with Cocktail substrate (Midazolam, dextromethorphan, Rosuvastatin and digoxin) on an empty stomach on Day 1. JMKX001899 was administered orally once daily after a standardized meal from Day 9 to Day 20 and Day 22. Cocktail and JMKX001899 were administered simultaneously on an empty stomach on Day 8 and Day 21.
  Interventions: Drug: JMKX001899; Drug: Midazolam; Drug: dextromethorphan; Drug: Rosuvastatin; Drug: digoxin

INTERVENTIONS:
Drug: JMKX001899 — Oral
Drug: Itraconazole — Oral
  Arms: JMKX001899+Itraconazole
Drug: Midazolam — Oral
  Arms: JMKX001899+Cocktail substrate (Midazolam, dextromethorphan, Rosuvastatin and digoxin)
Drug: Rifampin — Oral
  Arms: JMKX001899+Rifampin
Drug: dextromethorphan — Oral
  Arms: JMKX001899+Cocktail substrate (Midazolam, dextromethorphan, Rosuvastatin and digoxin)
Drug: Rosuvastatin — Oral
  Arms: JMKX001899+Cocktail substrate (Midazolam, dextromethorphan, Rosuvastatin and digoxin)
Drug: digoxin — Oral
  Arms: JMKX001899+Cocktail substrate (Midazolam, dextromethorphan, Rosuvastatin and digoxin)

SUMMARY:
This is an open-label, non-randomized, clinical study to evaluate the drug interaction between itraconazole, rifampin or Cocktail and JMKX001899 in healthy subjects. A total of three cohorts of 72 healthy subjects were planned to be enrolled in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily sign the informed consent, fully understand the content of the trial, and be able to complete the study according to the requirements of the trial protocol.
2. subjects aged 18 to 45 years (including both ends) at the time of signing informed consent.
3. male body weight is not less than 50 kg, female body weight is not less than 50 kg, and body mass index (BMI) is within the range of 19 ~ 27 kg/m2 (including cut-off value).

Exclusion Criteria:

1. hepatitis B surface antigen HBsAg positive, hepatitis C virus antibody positive, positive AIDS antigen/antibody or Treponema pallidum antibody.
2. Patients with a history of clinically significant diseases including, but not limited to, gastrointestinal, renal, liver, neurological, hematological, endocrine, neoplastic, pulmonary, immune, psychiatric, or cardiovascular and cerebrovascular diseases, epilepsy, bipolar disorder/mania, intraocular hypertension, or acute angle-closure glaucoma.
3. have taken any products containing caffeine, alcohol, grapefruit, and xanthine-rich within 24 hours before taking study medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
maximum concentrations (Cmax ) for plasma | approximately 3 days after first dose
area under the curve from time 0 to infinity(AUC0-inf) for plasma | approximately 3 days after first dose
area under the curve from time 0 to the last time point (AUC0-t) for plasma | approximately 3 days after first dose

IPD SHARING:
Plan to Share IPD: No